CLINICAL TRIAL: NCT04724785
Title: Real World Study on the Effect of HBV-DNA High-precision Detection Based Anti-viral Regimen Adjustment on Achieving Complete Virologic Response in Patients With Chronic Hepatitis B.(REACH)
Brief Title: Real World Study About Anti-viral Regimen Adjustment on Achieving Complete Response in CHB Patients
Acronym: REACH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, caidachuan, Dr/ Prof., The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2020LCYJ009
Record Dates: First submitted 2021-01-17; First posted 2021-01-26 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-01

CONDITIONS: Sustained Virologic Response; Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients with persistant low level HBV DNA (<10 IU/ml): No further intervention(s) to be administered except for monitoring of HBV DNA viraemia
  Interventions: Other: only monitoring
- patients with persistant HBV DNA (>10 IU/ml) but refuse to change the regimen: All patients with CHB receiving ETV or second-line NA(LAM/ADV/LdT) treatment for more than six months to one year will receive HBV-DNA detection, and patients with HBV-DNA≥10 IU/ml will be informed and recommended to adjust the treatment regimen. If those patients refuse to change the regimen which they are using , No further intervention(s) to be administered except for monitoring of HBV DNA viraemia until those patients change their idea
  Interventions: Other: monitoring and regimen change if necessary
- patients with persistant HBV DNA (>10 IU/ml) and agree to change the regimen: All patients with CHB receiving ETV or second-line NA(LAM/ADV/LdT) treatment for more than six months to one year will receive HBV-DNA detection, and patients with HBV-DNA≥10 IU/ml will be informed and recommended to adjust the treatment regimen.They will change their regimen according one which they are using.
  Interventions: Drug: regimen change

INTERVENTIONS:
Other: only monitoring — monitoring the viraemia only
  Groups: patients with persistant low level HBV DNA (<10 IU/ml)
Other: monitoring and regimen change if necessary — if those patients agree, the regimen will be changed.
  Groups: patients with persistant HBV DNA (>10 IU/ml) but refuse to change the regimen
Drug: regimen change — Based on ongoing one, regimen will be changed . The principle for adjusting anti-viral regimen is as follows: 1. The patients were treated with second-line drugs: changing ADV to ETV/TAF/TDF , changing LAM to TAF/TDF and changing LdT to TAF/TDF; 2. The patients were treated with ETV: adding or switching to TAF/TDF;3. TAF or ETV is recommended for patients with one or more TDF risk factors, such as > 40 years old, patients with abnormal bone/kidney related indicators or patients with high risk of bone/kidney injuries.【ADV=adefovir dipivoxil, LAM=lamivudine, and LdT=telbivudine , TAF =Tenofovir alafenamide Fumarate, ETV=Entecavir and TDF=Tenofovir disoproxil fumarate 】
  Groups: patients with persistant HBV DNA (>10 IU/ml) and agree to change the regimen

SUMMARY:
In the treatment of chronic hepatitis B (CHB), viral suppression is closely related to disease progression, and the lower the viral load, the lower the risk of progression to cirrhosis and hepatocellular carcinoma (HCC). In addition, a considerable number of patients in China are still using non-first-line antiviral therapy, such as adefovir dipivoxil, lamivudine, and telbivudine (ADV/LAM/LdT). About 25% of patients who received entecavir(ETV) treatment for more than half a year and confirmed that their DNA had turned negative by non-high-precision detection methods still had low viremia (LLV,DNA>20 IU/ml,IU=international unit), and LLV patients were twice as likely to develop HCC as patients with complete viral response.Patients who have received ETV or second-line NA(LAM/ADV/LdT) treatment for more than half a year to 1 year and confirmed HBV-DNA>10IU/ml by high-precision detection method are recommended to adjust the treatment plan in order to reduce the DNA load below 10IU/ml as soon as possible. It is up to the doctor, in consultation with the patient, to decide whether or not to make the adjustment.

DETAILED DESCRIPTION:
In our hospital, about 150 patients are screened for HBV-DNA every day. Therefore, 54 million patients will be tested for HBV-DNA within one year, of which 30% are estimated to be HBV-DNA ≥10 IU. These patients will be informed to the Department of Infectious Diseases of the Second Affiliated Hospital of Chongqing Medical University for follow-up, and will be randomly divided into three groups according to 1:1. Patients in all three groups will be educated about hepatitis B virus infection and antiviral treatment, and the treatment regimen will be adjusted according to whether their HBV DNA is ≥10 IU/ml or not. Patients in group 1: patients with persistant low level HBV DNA (<10 IU/ml). Patients in group 2: HBV-DNA≥10 IU/ml, receiving HBV-related education and being advised by the doctor to change or to add another NA. Patients in group 2: patients with persistant HBV DNA (>10 IU/ml) but refuse to change the regimen. Patients in group 3: patients with persistant HBV DNA (>10 IU/ml) and agree to change the regimen. Educational methods include videos, including an introduction to hepatitis B virus (disease profile, infection, outcome, HBV infection, vertical transmission and other risk factors) for 5 minutes, brochures with relevant information and consultations with physicians and nurses.

All patients with chronic hepatitis B(CHB) receiving ETV or second-line NA(LAM/ADV/LdT) treatment for more than six months to one year will receive HBV-DNA detection, and patients with HBV-DNA≥10 IU/ml will be informed and recommended to adjust the treatment regimen so that the actual prevalence of HBV-DNA load < 10 IU/ml in Chongqing HBV cohort could be obtained . The investigators estimated that 30% of the patients had HBV-DNA≥ 10 IU/ml, so there were about 16,200 patients had HBV-DNA≥ 10 IU/ml among 54,000 patients a year. These patients will be diagnosed with LLV and will undergo a treatment regimen adjustment, with a recommendation to switch to or use a different type of nucleos(t)ide analogue (NA) for anti-viral treatment.

ELIGIBILITY:
Inclusion Criteria:

* any patients treated with ETV\LAM\ADF\LDT\TDF\TAF.【ADV=adefovir dipivoxil, LAM=lamivudine, and LdT=telbivudine , TAF =Tenofovir alafenamide Fumarate, ETV=Entecavir and TDF=Tenofovir disoproxil fumarate 】

Exclusion Criteria:

* with a expected life span <48 weeks

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research subjects were patients with CHB (chronic hepatitis B) receiving ETV or second-line NA(LAM/ADV/LdT) who were admitted to The Second Affiliated Hospital of Chongqing Medical University and other centers.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who received a complete virologic response (HBV DNA<10IU/ml) at 24 weeks after therapy adjustment. | 24 weeks
  The proportion of patients who received a complete virologic response (HBV DNA<10IU/ml) at 24 weeks after therapy adjustment.

SECONDARY OUTCOMES:
The proportion of patients with complete virologic response (HBV DNA<10IU/ml) at 12 weeks, 48 weeks and 96 weeks after therapy adjustment. | 12 weeks, 48 weeks ,96 weeks
  The proportion of patients with complete virologic response (HBV DNA<10IU/ml) at 12 weeks, 48 weeks and 96 weeks after therapy adjustment.
he proportion of patients with normal Alanine transaminase（ALT） at baseline and at each follow-up time point | baseline,12 weeks,48 weeks,96 weeks
  he proportion of patients with normal Alanine transaminase（ALT ）at baseline and at each follow-up time point
Changes of estimated glomerularfiltrationratee(GFR) compared with baseline at each follow-up time point. | baseline,12 weeks,48 weeks,96 weeks
  Changes of estimated glomerularfiltrationratee(GFR) compared with baseline at each follow-up time point.
Changes of serum creatinine(SCr）compared with baseline at each follow-up time point. | baseline,12 weeks,48 weeks,96 weeks
  Changes of serum creatinine(SCr) compared with baseline at each follow-up time point.
Changes of bone mass density（BMD) compared with baseline at each follow-up time point. | baseline,12 weeks,48 weeks,96 weeks
  Changes of bone mass density (BMD) compared with baseline at each follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: DACHUAN CAI, PhD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The second affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui F, Shen L, Li L, Wang H, Wang F, Bi S, Liu J, Zhang G, Wang F, Zheng H, Sun X, Miao N, Yin Z, Feng Z, Liang X, Wang Y. Prevention of Chronic Hepatitis B after 3 Decades of Escalating Vaccination Policy, China. Emerg Infect Dis. 2017 May;23(5):765-772. doi: 10.3201/eid2305.161477. PMID 28418296
- [Background] Liu J, Liang W, Jing W, Liu M. Countdown to 2030: eliminating hepatitis B disease, China. Bull World Health Organ. 2019 Mar 1;97(3):230-238. doi: 10.2471/BLT.18.219469. Epub 2019 Jan 28. PMID 30992636
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Chen JD, Yang HI, Iloeje UH, You SL, Lu SN, Wang LY, Su J, Sun CA, Liaw YF, Chen CJ; Risk Evaluation of Viral Load Elevation and Associated Liver Disease/Cancer in HBV (REVEAL-HBV) Study Group. Carriers of inactive hepatitis B virus are still at risk for hepatocellular carcinoma and liver-related death. Gastroenterology. 2010 May;138(5):1747-54. doi: 10.1053/j.gastro.2010.01.042. Epub 2010 Jan 28. PMID 20114048
- [Background] Liu C, Wang L, Xie H, Zhang L, Wang B, Luo C, Wang S, Tang M, Fu Z, Ruan H, Liu Z, Wei L, Yi W, Xie Y. The relationship between serum hepatitis B virus DNA level and liver histology in patients with chronic HBV infection. PLoS One. 2018 Nov 7;13(11):e0206060. doi: 10.1371/journal.pone.0206060. eCollection 2018. PMID 30403735
- [Background] Zhang W, Wang X, Wang Y, Zhao X, Duan W, Wang Q, Wu X, Kong Y, Ma H, You H, Ou X, Jia J. Effective viral suppression is necessary to reduce hepatocellular carcinoma development in cirrhotic patients with chronic hepatitis B: Results of a 10-year follow up. Medicine (Baltimore). 2017 Nov;96(44):e8454. doi: 10.1097/MD.0000000000008454. PMID 29095292
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Ogawa E, Nomura H, Nakamuta M, Furusyo N, Koyanagi T, Dohmen K, Ooho A, Satoh T, Kawano A, Kajiwara E, Takahashi K, Azuma K, Kato M, Shimoda S, Hayashi J; Kyushu University Liver Disease Study (KULDS) Group. Tenofovir alafenamide after switching from entecavir or nucleos(t)ide combination therapy for patients with chronic hepatitis B. Liver Int. 2020 Jul;40(7):1578-1589. doi: 10.1111/liv.14482. Epub 2020 Apr 30. PMID 32304611
- [Background] Sun Y, Wu X, Zhou J, Meng T, Wang B, Chen S, Liu H, Wang T, Zhao X, Wu S, Kong Y, Ou X, Wee A, Theise ND, Qiu C, Zhang W, Lu F, Jia J, You H. Persistent Low Level of Hepatitis B Virus Promotes Fibrosis Progression During Therapy. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2582-2591.e6. doi: 10.1016/j.cgh.2020.03.001. Epub 2020 Mar 6. PMID 32147592
- [Background] Kim JH, Sinn DH, Kang W, Gwak GY, Paik YH, Choi MS, Lee JH, Koh KC, Paik SW. Low-level viremia and the increased risk of hepatocellular carcinoma in patients receiving entecavir treatment. Hepatology. 2017 Aug;66(2):335-343. doi: 10.1002/hep.28916. Epub 2016 Dec 24. PMID 28012257
- [Background] Jang JW, Choi JY, Kim YS, Yoo JJ, Woo HY, Choi SK, Jun CH, Lee CH, Sohn JH, Tak WY, Lee YR, Han KH. Effects of Virologic Response to Treatment on Short- and Long-term Outcomes of Patients With Chronic Hepatitis B Virus Infection and Decompensated Cirrhosis. Clin Gastroenterol Hepatol. 2018 Dec;16(12):1954-1963.e3. doi: 10.1016/j.cgh.2018.04.063. Epub 2018 May 9. PMID 29753085
- [Background] Wang J, Sheng Q, Ding Y, Chen R, Sun X, Chen X, Dou X, Lu F. HBV RNA virion-like particles produced under nucleos(t)ide analogues treatment are mainly replication-deficient. J Hepatol. 2018 Apr;68(4):847-849. doi: 10.1016/j.jhep.2017.10.030. Epub 2017 Nov 4. No abstract available. PMID 29113914
- [Background] Dandri M, Petersen J. Mechanism of Hepatitis B Virus Persistence in Hepatocytes and Its Carcinogenic Potential. Clin Infect Dis. 2016 Jun 1;62 Suppl 4(Suppl 4):S281-8. doi: 10.1093/cid/ciw023. PMID 27190317
- [Background] Kim HJ, Cho YK, Jeon WK, Kim BI. Clinical characteristics of patients with chronic hepatitis B who developed genotypic resistance to entecavir: Real-life experience. Clin Mol Hepatol. 2017 Dec;23(4):323-330. doi: 10.3350/cmh.2017.0005. Epub 2017 Sep 5. PMID 28870025
- [Background] Wong GL, Wong VW, Chan HY, Tse PC, Wong J, Chim AM, Yiu KK, Chu SH, Chan HL. Undetectable HBV DNA at month 12 of entecavir treatment predicts maintained viral suppression and HBeAg-seroconversion in chronic hepatitis B patients at 3 years. Aliment Pharmacol Ther. 2012 Jun;35(11):1326-35. doi: 10.1111/j.1365-2036.2012.05098.x. Epub 2012 Apr 16. PMID 22506552
- [Background] Sun Y, Zhou J, Wang L, Wu X, Chen Y, Piao H, Lu L, Jiang W, Xu Y, Feng B, Nan Y, Xie W, Chen G, Zheng H, Li H, Ding H, Liu H, Lv F, Shao C, Wang T, Ou X, Wang B, Chen S, Wee A, Theise ND, You H, Jia J. New classification of liver biopsy assessment for fibrosis in chronic hepatitis B patients before and after treatment. Hepatology. 2017 May;65(5):1438-1450. doi: 10.1002/hep.29009. Epub 2017 Mar 22. PMID 28027574
- [Background] Yenilmez E, Cetinkaya RA, Tural E. Diagnostic Dilemma for Low Viremia with Significant Fibrosis; is Hepatitis B Virus DNA Threshold Level a Good Indicator for Predicting Liver Damage? Balkan Med J. 2018 Jul 24;35(4):326-332. doi: 10.4274/balkanmedj.2017.0888. Epub 2018 May 4. PMID 29726399
- [Background] Sinn DH, Lee J, Goo J, Kim K, Gwak GY, Paik YH, Choi MS, Lee JH, Koh KC, Yoo BC, Paik SW. Hepatocellular carcinoma risk in chronic hepatitis B virus-infected compensated cirrhosis patients with low viral load. Hepatology. 2015 Sep;62(3):694-701. doi: 10.1002/hep.27889. Epub 2015 Jul 3. PMID 25963803
- [Background] Papatheodoridis GV, Manolakopoulos S, Touloumi G, Vourli G, Raptopoulou-Gigi M, Vafiadis-Zoumbouli I, Vasiliadis T, Mimidis K, Gogos C, Ketikoglou I, Manesis EK; HEPNET. Greece Cohort Study Group. Virological suppression does not prevent the development of hepatocellular carcinoma in HBeAg-negative chronic hepatitis B patients with cirrhosis receiving oral antiviral(s) starting with lamivudine monotherapy: results of the nationwide HEPNET. Greece cohort study. Gut. 2011 Aug;60(8):1109-16. doi: 10.1136/gut.2010.221846. Epub 2011 Jan 26. PMID 21270118
- [Background] Nam JY, Chang Y, Cho H, Kang SH, Cho YY, Cho EJ, Lee JH, Yu SJ, Yoon JH, Kim YJ. Delayed viral suppression during antiviral therapy is associated with increased hepatocellular carcinoma rates in HBeAg-positive high viral load chronic hepatitis B. J Viral Hepat. 2018 May;25(5):552-560. doi: 10.1111/jvh.12838. Epub 2018 Mar 14. PMID 29194870
- [Background] Kim TS, Sinn DH, Kang W, Gwak GY, Paik YH, Choi MS, Lee JH, Koh KC, Paik SW. Hepatitis B virus DNA levels and overall survival in hepatitis B-related hepatocellular carcinoma patients with low-level viremia. J Gastroenterol Hepatol. 2019 Nov;34(11):2028-2035. doi: 10.1111/jgh.14750. Epub 2019 Jul 28. PMID 31157456
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] Korean Association for the Study of the Liver. KASL Clinical Practice Guidelines: Management of chronic hepatitis B. Clin Mol Hepatol. 2012 Jun;18(2):109-62. doi: 10.3350/cmh.2012.18.2.109. Epub 2012 Jun 26. PMID 22893865
- [Background] Yim HJ, Kim IH, Suh SJ, Jung YK, Kim JH, Seo YS, Yeon JE, Kim CW, Kwon SY, Park SH, Lee MS, Um SH, Byun KS. Switching to tenofovir vs continuing entecavir for hepatitis B virus with partial virologic response to entecavir: a randomized controlled trial. J Viral Hepat. 2018 Nov;25(11):1321-1330. doi: 10.1111/jvh.12934. Epub 2018 Jun 6. PMID 29772084
- [Background] Lu L, Yip B, Trinh H, Pan CQ, Han SH, Wong CC, Li J, Chan S, Krishnan G, Wong CC, Nguyen MH. Tenofovir-based alternate therapies for chronic hepatitis B patients with partial virological response to entecavir. J Viral Hepat. 2015 Aug;22(8):675-81. doi: 10.1111/jvh.12368. Epub 2014 Nov 24. PMID 25417914
- [Background] Lim YS, Yoo BC, Byun KS, Kwon SY, Kim YJ, An J, Lee HC, Lee YS. Tenofovir monotherapy versus tenofovir and entecavir combination therapy in adefovir-resistant chronic hepatitis B patients with multiple drug failure: results of a randomised trial. Gut. 2016 Jun;65(6):1042-51. doi: 10.1136/gutjnl-2014-308435. Epub 2015 Mar 23. PMID 25800784
- [Background] Chen J, Zhao SS, Liu XX, Huang ZB, Huang Y. Comparison of the Efficacy of Tenofovir Versus Tenofovir plus Entecavir in the Treatment of Chronic Hepatitis B in Patients With Poor Efficacy of Entecavir: A Systematic Review and Meta-analysis. Clin Ther. 2017 Sep;39(9):1870-1880. doi: 10.1016/j.clinthera.2017.07.015. Epub 2017 Aug 7. PMID 28797777
- [Background] Wang YH, Liao J, Zhang DM, Wu DB, Tao YC, Wang ML, Chen EQ, Tang H. Tenofovir monotherapy versus tenofovir plus entecavir combination therapy in HBeAg-positive chronic hepatitis patients with partial virological response to entecavir. J Med Virol. 2020 Mar;92(3):302-308. doi: 10.1002/jmv.25608. Epub 2019 Oct 29. PMID 31609007

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04724785/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04724785/ICF_001.pdf